CLINICAL TRIAL: NCT03492645
Title: Technology and Telephone-Based Smoking Cessation Treatment for Veterans With Posttraumatic Stress Disorder
Brief Title: Technology and Telephone-Based Smoking Cessation
Acronym: RAP Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-21605
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Office Group (Active Comparator)
  Interventions: Behavioral: Office-based treatment protocol
- Telephone Group (Experimental)
  Interventions: Behavioral: Telephone-and technology-facilitated treatment protocol

INTERVENTIONS:
Behavioral: Telephone-and technology-facilitated treatment protocol — 1. 8 video or telephone counseling sessions targeting PTSD symptoms related to smoking lapse. The first of these sessions will last approximately 45-60 minutes, and the remaining 7 sessions will last 20-30 minutes.
  2. Use of the Stay Quit Coach (SQC) app between sessions. SQC is a public domain, no-cost mobile app designed by our co-investigators at the National Center for PTSD to complement the IC protocol with evidence-based tools to support smoking cessation, such as motivational messaging and coping tools for managing PTSD symptoms associated with smoking lapse.
  3. Use of the Covita Bedfont iCO Smokerlyzer, a mobile carbon monoxide (CO) monitor, compatible with iOS and Android smartphones, that provides CO readings to the user at any time in order to self-monitor progress in quitting. The Covita iCO mobile app is used with the iCO Smoerlyzer to display CO readings.
  Arms: Telephone Group
Behavioral: Office-based treatment protocol — Weekly face-to-face sessions using the unmodified treatment manual developed by McFall and Saxon, a protocol combining office-based therapy plus evidence-based pharmacotherapies for smoking cessation that doubled quit rates in veteran smokers with PTSD.
  Arms: Office Group

SUMMARY:
The goal of the proposed project is to design and assess the acceptability and usability of a mobile technology and telephone-facilitated treatment to improve treatment engagement in adult smokers with posttraumatic stress disorder (PTSD). Smokers with PTSD face high rates of treatment failure and require tailored strategies that address both PTSD symptoms and smoking urges. McFall and Saxon designed a protocol combining office-based therapy plus evidence-based pharmacotherapies for smoking cessation that doubled quit rates in veteran smokers with PTSD. However, high rates of attrition limited efficacy. The investigators aim to enhance scalability and engagement in the McFall/ Saxon protocol by (1) adapting the treatment to be delivered over the video or telephone and (2) leveraging innovations in technology by incorporating a mobile application targeting PTSD and smoking and a mobile carbon monoxide (CO) monitor into the protocol. The investigators propose a mixed methods study in which the investigators will adapt the office-based treatment into a technology and telephone-facilitated intervention and conduct a pilot RCT of the modified intervention with 20 veterans with PTSD. At the outset of the study, the study team will modify the original treatment manual in order for it to be delivered via video or telephone. The investigators will then conduct a pilot RCT in which 20 veterans with PTSD will be randomized to receive the modified protocol (intervention condition; n=10) or the original office-based protocol (control condition, n=10). Main outcomes are quantitative and qualitative data about the acceptability of the intervention and its individual components, and treatment retention at Week 8. Secondary outcomes are 7-day bioverified point-prevalence cigarette abstinence, PTSD symptoms, and levels of nicotine dependence at follow-up. Results will inform a larger RCT to examine efficacy of the intervention in promoting quit attempts in smokers with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* are a veteran ages 18-69 meeting lifetime criteria for PTSD using the Diagnostic Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) as assessed by the MINI International Neuropsychiatric Interview
* have smoked at least five cigarettes per day on at least 15 of 30 days before screening
* are interested in smoking cessation
* are willing to receive smoking cessation interventions
* are a smartphone (iOS or Android) user

Exclusion Criteria:

* women who are pregnant or plan to become pregnant
* current and unstable psychotic or bipolar disorder (potential participants whose symptoms are treated and stable may participate)
* current severe psychiatric symptoms or psychiatric instability
* current severe substance use disorder
* cognitive impairment assessed by Montreal Cognitive Assessment (MoCA) Score below 23

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) for iCO monitor and Stay Quit Coach (SQC) App | Week 8
  The SUS is a brief, reliable and valid instrument to measure perceptions of usability of technology devices. Items are rated on a scale from 0-5. An SUS total score is calculated by summing item ratings, and then multiplied the sum by 2.5. The maximum score on the SUS is 100, with higher scores reflecting greater usability. We will administer the SUS to the intervention condition only. Mean usability score will be reported.
Acceptability questionnaire | Week 8
  Participants (in the intervention condition only) will complete a questionnaire developed by our team to rate the intervention protocol from 1-10 in terms of perceived helpfulness, understandability, and likelihood of use. The mean score (i.e., average of item ratings) will be reported for the participants in the intervention condition. Higher scores represent greater acceptability.
Client Satisfaction Questionnaire-8 | Week 8
  The CSQ-8 is an eight-item instrument designed to measure satisfaction with an clinical intervention. Items are rated on a scale from 1-4 and summed to for an CSQ-8 total score. Scores range from 8-32, with higher scores indicating greater satisfaction. We will administer the CSQ-8 to the intervention condition only. Mean satisfaction score will be reported.
Total number of treatment sessions completed | Week 1-8
  We will record attendance at each session Weeks 1-8 in both arms.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-5) | Weeks 0 & 8
  The PCL-5 is a 20-item self-report measure that assesses the severity of the twenty DSM-V symptoms of PTSD. Items are rated on a 1-5 scale and summed to compute a total score, with higher scores representing greater severity of PTSD symptoms. This outcome variable will be reported as the difference in PCL-5 total score between the experimental treatment condition and the control condition.
Number of cigarettes smoked | Weeks 0 & 8
  Self-reported use of cigarettes will be assessed with TLFB (past 30 days), which uses a calendar with specific anchor dates to identify the quantity and frequency of use. This outcome variable will be reported as the difference in cigarette use between the experimental treatment condition and the control condition.
Carbon monoxide levels | Weeks 0 & 8
  Exhaled CO will be obtained in person with a Covita office Smokerlyzer
Fagerstrom Test of Nicotine Dependence (FTND) scores | Weeks 0 & 8
  The FTND is a validated, 6-item self-report instrument that evaluates the intensity of physical addiction to nicotine. Three items are rated yes/no (0/1), and the other three items are rated on a scale from 0-3. Items are summed to yield a total score of 0-10, with higher scores reflecting greater nicotine dependence. This outcome variable will be reported as the difference in FTND total score between the experimental treatment condition and the control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States